CLINICAL TRIAL: NCT03522506
Title: A Phase 1b, 4-Period Crossover, Placebo-Controlled, Randomized, Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAK-925 in Sleep-Deprived Healthy Adults Utilizing Modafinil as an Active Comparator
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of TAK-925 Study in Sleep-Deprived Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-925-1002; U1111-1211-2133 (Other: WHO)
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Results first posted 2019-11-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-925; Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TAK-925 Low Dose + Placebo + TAK-925 High Dose + Modafinil (Experimental): TAK-925 low dose milligram (mg), intravenously, administered as 9-hour infusion, once on Day 1 of Intervention Period 1, followed by a minimum of 7-days washout period, further followed by placebo once on Day 1 of Intervention Period 2, followed by a minimum of 7-days washout period, further followed by TAK-925 high dose mg, intravenously, administered as 9-hour infusion, once on Day 1 of Intervention Period 3, followed by a minimum of 7-days washout period, further followed by Modafinil 300 mg, tablet, orally, once on Day 1 of Intervention Period 4. TAK-925 dose will be decided based on the availability of safety, tolerability and PK data from ongoing study TAK-925-1001.
  Interventions: Drug: TAK-925; Drug: TAK-925 Placebo; Drug: Modafinil; Drug: Modafinil Placebo
- TAK-925 High Dose + TAK-925 Low Dose + Modafinil + Placebo (Experimental): TAK-925 high dose mg, intravenously, administered as 9-hour infusion, once on Day 1 of Intervention Period 1, followed by a minimum of 7-days washout period, further followed by TAK-925 low dose mg, intravenously, administered as 9-hour infusion, once on Day 1 of Intervention Period 2, followed by a minimum of 7-days washout period, further followed by Modafinil 300 mg, tablet, orally, once on Day 1 of Intervention Period 3, followed by a minimum of 7-days washout period, further followed by placebo once on Day 1 of Intervention Period 4. TAK-925 dose will be decided based on the availability of safety, tolerability and PK data from ongoing study TAK-925-1001.
  Interventions: Drug: TAK-925; Drug: TAK-925 Placebo; Drug: Modafinil; Drug: Modafinil Placebo
- Modafinil + TAK-925 High Dose + Placebo + TAK-925 Low Dose (Experimental): Modafinil 300 mg, tablet, orally, once on Day 1 of Intervention Period 1, followed by a minimum of 7-days washout period, further followed by TAK-925 high dose mg, intravenously, administered as 9-hour infusion, once on Day 1 of Intervention Period 2, followed by a minimum of 7-days washout period, further followed by placebo once on Day 1 of Intervention Period 3, followed by a minimum of 7-days washout period, further followed by TAK-925 low dose mg, intravenously, administered as 9-hour infusion, once on Day 1 of Intervention Period 4. TAK-925 dose will be decided based on the availability of safety, tolerability and PK data from ongoing study TAK-925-1001.
  Interventions: Drug: TAK-925; Drug: TAK-925 Placebo; Drug: Modafinil; Drug: Modafinil Placebo
- Placebo + Modafinil + TAK-925 Low Dose + TAK-925 High Dose (Experimental): Placebo, once on Day 1 of Intervention Period 1, followed by a minimum of 7-days washout period, further followed by Modafinil 300 mg, tablet, orally, once on Day 1 of Intervention Period 2, followed by a minimum of 7-days washout period, further followed by TAK-925 low dose mg, intravenously, administered as 9-hour infusion, once on Day 1 of Intervention Period 3, followed by a minimum of 7-days washout period, further followed by TAK-925 high dose mg, intravenously, administered as 9-hour infusion, once on Day 1 of Intervention Period 4. TAK-925 dose will be decided based on the availability of safety, tolerability and PK data from ongoing study TAK-925-1001.
  Interventions: Drug: TAK-925; Drug: TAK-925 Placebo; Drug: Modafinil; Drug: Modafinil Placebo

INTERVENTIONS:
Drug: TAK-925 — TAK-925 intravenous infusion.
Drug: TAK-925 Placebo — TAK-925 placebo-matching given as saline intravenous infusion.
Drug: Modafinil — Modafinil tablets.
Drug: Modafinil Placebo — Modafinil placebo-matching tablet.

SUMMARY:
The purpose of this study is to determine the effect of TAK-925 after a single intravenous dose (compared to placebo) on promoting wakefulness as measured by sleep latency on the maintenance of wakefulness (MWT) in sleep-deprived healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-925. This study will assess the safety, tolerability, PK and PD of TAK-925 and will assess the effects of TAK-925 in sleep-deprived healthy adult participants.

The study will enroll approximately 20 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the 4 treatment sequences-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-925 Low Dose + Placebo + TAK-925 High Dose + Modafinil
* TAK-925 High Dose + TAK-925 Low Dose + Modafinil + Placebo
* Modafinil+ TAK-925 High Dose + Placebo + TAK-925 Low Dose
* Placebo + Modafinil + TAK-925 Low Dose + TAK-925 High Dose

TAK-925 will be administered as an intravenous infusion based on the availability of safety, tolerability and PK data from health Japanese participants in ongoing study TAK-925-1001.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 10 weeks. Participants will make a final visit 7 days after receiving their last dose of drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Be a nonsmoker who has not used tobacco- or nicotine-containing products (example, nicotine patch) for at least 6 months before study drug administration of the initial dose of study drug.
2. Have regular sleep-wake habits (example, routinely spending 6.5 to 8 hours sleeping nightly, not oversleeping by more than 3 hours on weekends, that is, total sleep not more than 11 hours) as determined by investigator interviews and confirmed in 5-day actigraphy records and whom regularly fall asleep between 9:30 PM and 12:00 AM.
3. Be willing to have actigraphy monitoring during the week before randomization and in each interval.

Exclusion Criteria:

1. Has a positive alcohol or drug screen.
2. Has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to: beer [354 milliliter per (mL/)12 ounces], wine (118 mL/4 ounces), or distilled spirits (29.5 mL/1 ounce)] per day).
3. Has excessive sleepiness defined by a self-reported Epworth Sleepiness Scale score at screening greater than 10; irregular work hours; or routine night-shift work within 1 month before randomization.
4. Currently experiencing or having a history of any known/suspected sleep disorder, any disorder associated with excessive daytime somnolence (EDS), or any diagnosis interfering with assessment of sleepiness.
5. Abnormal findings on the initial polysomnography (PSG) conducted on Day -1 (check-in), as specified in the study manual.
6. Traveled across 2 or more time zones 2 weeks or less before screening.
7. Caffeine consumption of more than 400 milligram per day (mg/day) for 2 weeks before screening (1 serving of coffee is approximately equivalent to 120 mg of caffeine).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Evans R, Kimura H, Nakashima M, Ishikawa T, Yukitake H, Suzuki M, Hazel J, Faessel H, Wu J, Hang Y, Alexander R, Rosen L, Hartman DS, Ratti E. Orexin 2 receptor-selective agonist danavorexton (TAK-925) promotes wakefulness in non-human primates and healthy individuals. J Sleep Res. 2023 Oct;32(5):e13878. doi: 10.1111/jsr.13878. Epub 2023 Mar 19. PMID 36934366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 09 May 2018 to 07 November 2018.
Pre-assignment Details: Healthy sleep deprived participants were enrolled in 1 of the 4 treatment sequences of this 4-period crossover study to receive: TAK 925 44 milligram (mg) (Low dose), TAK-925 112 mg (High dose), modafinil 300 mg, and placebo.
Groups:
- TAK-925 44 mg + Placebo + TAK-925 112 mg + Modafinil 300 mg: TAK-925 44 mg, injection, intravenously, administered as 9-hour infusion, once on Day 1 of Treatment Period 1, followed by a minimum of 7-days washout period, further followed by placebo once on Day 1 of Treatment Period 2, followed by a minimum of 7-days washout period, further followed by TAK-925 112 mg, injection, intravenously, administered as 9-hour infusion, once on Day 1 of Treatment Period 3, followed by a minimum of 7-days washout period, further followed by modafinil 300 mg, tablet, orally, once on Day 1 of Treatment Period 4.
- TAK-925 112 mg + TAK-925 44 mg + Modafinil 300 mg + Placebo: TAK-925 112 mg, injection, intravenously, administered as 9-hour infusion, once on Day 1 of Treatment Period 1, followed by a minimum of 7-days washout period, further followed by TAK-925 44 mg, injection, intravenously, administered as 9-hour infusion, once on Day 1 of Treatment Period 2, followed by a minimum of 7-days washout period, further followed by modafinil 300 mg, tablet, orally, once on Day 1 of Treatment Period 3, followed by a minimum of 7-days washout period, further followed by placebo once on Day 1 of Treatment Period 4.
- Modafinil 300 mg + TAK-925 112 mg + Placebo + TAK-925 44 mg: Modafinil 300 mg, tablet, orally, once on Day 1 of Treatment Period 1, followed by a minimum of 7-days washout period, further followed by TAK-925 112 mg, injection, intravenously, administered as 9-hour infusion, once on Day 1 of Treatment Period 2, followed by a minimum of 7-days washout period, further followed by placebo once on Day 1 of Treatment Period 3, followed by a minimum of 7-days washout period, further followed by TAK-925 44 mg, injection, intravenously, administered as 9-hour infusion, once on Day 1 of Treatment Period 4.
- Placebo + Modafinil 300 mg + TAK-925 44 mg + TAK-925 112 mg: Placebo, once on Day 1 of Treatment Period 1, followed by a minimum of 7-days washout period, further followed by modafinil 300 mg, tablet, orally, once on Day 1 of Treatment Period 2, followed by a minimum of 7-days washout period, further followed by TAK-925 44 mg, injection, intravenously, administered as 9-hour infusion, once on Day 1 of Treatment Period 3, followed by a minimum of 7-days washout period, further followed by TAK-925 112 mg, injection, intravenously, administered as 9-hour infusion, once on Day 1 of Treatment Period 4.
Period: Treatment Period 1 (2 Days)
Arm/Group | TAK-925 44 mg + Placebo + TAK-925 112 mg + Modafinil 300 mg | TAK-925 112 mg + TAK-925 44 mg + Modafinil 300 mg + Placebo | Modafinil 300 mg + TAK-925 112 mg + Placebo + TAK-925 44 mg | Placebo + Modafinil 300 mg + TAK-925 44 mg + TAK-925 112 mg
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | TAK-925 44 mg + Placebo + TAK-925 112 mg + Modafinil 300 mg | TAK-925 112 mg + TAK-925 44 mg + Modafinil 300 mg + Placebo | Modafinil 300 mg + TAK-925 112 mg + Placebo + TAK-925 44 mg | Placebo + Modafinil 300 mg + TAK-925 44 mg + TAK-925 112 mg
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Treatment Period 2 (2 Days)
Arm/Group | TAK-925 44 mg + Placebo + TAK-925 112 mg + Modafinil 300 mg | TAK-925 112 mg + TAK-925 44 mg + Modafinil 300 mg + Placebo | Modafinil 300 mg + TAK-925 112 mg + Placebo + TAK-925 44 mg | Placebo + Modafinil 300 mg + TAK-925 44 mg + TAK-925 112 mg
Started | 5 | 5 | 5 | 4
Completed | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | TAK-925 44 mg + Placebo + TAK-925 112 mg + Modafinil 300 mg | TAK-925 112 mg + TAK-925 44 mg + Modafinil 300 mg + Placebo | Modafinil 300 mg + TAK-925 112 mg + Placebo + TAK-925 44 mg | Placebo + Modafinil 300 mg + TAK-925 44 mg + TAK-925 112 mg
Started | 5 | 5 | 5 | 4
Completed | 5 | 5 | 5 | 3
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Treatment Period 3 (2 Days)
Arm/Group | TAK-925 44 mg + Placebo + TAK-925 112 mg + Modafinil 300 mg | TAK-925 112 mg + TAK-925 44 mg + Modafinil 300 mg + Placebo | Modafinil 300 mg + TAK-925 112 mg + Placebo + TAK-925 44 mg | Placebo + Modafinil 300 mg + TAK-925 44 mg + TAK-925 112 mg
Started | 5 | 5 | 5 | 3
Completed | 5 | 5 | 5 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3 (7 Days)
Arm/Group | TAK-925 44 mg + Placebo + TAK-925 112 mg + Modafinil 300 mg | TAK-925 112 mg + TAK-925 44 mg + Modafinil 300 mg + Placebo | Modafinil 300 mg + TAK-925 112 mg + Placebo + TAK-925 44 mg | Placebo + Modafinil 300 mg + TAK-925 44 mg + TAK-925 112 mg
Started | 5 | 5 | 5 | 3
Completed | 5 | 5 | 5 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4 (2 Days)
Arm/Group | TAK-925 44 mg + Placebo + TAK-925 112 mg + Modafinil 300 mg | TAK-925 112 mg + TAK-925 44 mg + Modafinil 300 mg + Placebo | Modafinil 300 mg + TAK-925 112 mg + Placebo + TAK-925 44 mg | Placebo + Modafinil 300 mg + TAK-925 44 mg + TAK-925 112 mg
Started | 5 | 5 | 5 | 3
Completed | 5 | 5 | 5 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-925 44 mg + Placebo + TAK-925 112 mg + Modafinil 300 mg | TAK-925 112 mg + TAK-925 44 mg + Modafinil 300 mg + Placebo | Modafinil 300 mg + TAK-925 112 mg + Placebo + TAK-925 44 mg | Placebo + Modafinil 300 mg + TAK-925 44 mg + TAK-925 112 mg | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (4.55) | 26.4 (3.78) | 27.4 (3.44) | 26.0 (1.22) | 26.9 (3.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 3 | 7
  Not Hispanic or Latino | 4 | 5 | 2 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 5 | 5 | 4 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 5 | 5 | 20
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 82.6 (11.10) | 78.8 (6.52) | 84.2 (10.73) | 83.0 (11.59) | 82.2 (9.58)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 182.1 (5.32) | 176.1 (5.83) | 175.6 (8.60) | 175.2 (4.70) | 177.3 (6.46)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.9 (2.95) | 25.4 (1.31) | 27.2 (1.67) | 27.0 (2.89) | 26.1 (2.36)

OUTCOME MEASURES:

1. Primary Outcome: Latency to Sleep Onset on Maintenance of Wakefulness Test (MWT) at 2 Hours Post-infusion Start
Description: The MWT is a validated objective measure that evaluates a person's ability to remain awake under soporific conditions for a defined period of time. This tendency to fall asleep is measured via electroencephalography-derived sleep latency. Sleep onset is defined as the first epoch of greater than 15 seconds of cumulative sleep in a 30-second epoch. Trials were ended after 40 minutes if no sleep occurs, or after unequivocal sleep, defined as 3 consecutive epochs of stage 1 sleep, or 1 epoch of any other stage of sleep. If no sleep has been observed according to these rules, then the latency is defined as 40 minutes. MWT sleep latency ranges from 0 to 40 minutes, with higher scores indicating greater ability to stay awake.
Time Frame: Day 1: 2 hours post-infusion start
Population: Pharmacodynamics (PD) analysis set: all participants who received at least 1 dose of study drug and have at least 1 evaluable postdose PD endpoint derived from MWT, polysomnography (PSG), Karolinska Sleepiness Scale (KSS), or Cambridge Cognition Computerized Battery of Tests (CCBT). PD analysis set where data at specified time points was available.
Measure: Least Squares Mean (Standard Error); unit: minute
Groups:
- Placebo: Placebo, once on Day 1 of Treatment Period 1, 2, 3, or 4.
- TAK-925 44 mg: TAK-925 44 mg, intravenously, injection, administered as 9-hour infusion, once on Day 1 of Treatment Period 1, 2, 3, or 4.
- TAK-925 112 mg: TAK-925 112 mg, intravenously, injection, administered as 9-hour infusion, once on Day 1 of Treatment Period 1, 2, 3, or 4.
- Modafinil 300 mg: Modafinil 300 mg, tablet, orally, once on Day 1 of Treatment Period 1, 2, 3, or 4.
Arm/Group | Placebo | TAK-925 44 mg | TAK-925 112 mg | Modafinil 300 mg
Number analyzed (Participants) | 20 | 18 | 18 | 19
minute | 15.68 (2.305) | 35.74 (2.445) | 40.02 (2.445) | 35.57 (2.368)
Statistical Analysis 1: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — The effect of TAK-925 was evaluated with a linear mixed effects model appropriate for a 4-period crossover study. The least squares mean (LSM) sleep latency for each treatment and the associated standard error and 95% confidence interval (CI) was estimated from the model at each time, along with differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p < 0.001, Linear mixed effect model; Least square mean difference = 20.06, 95% CI 2-sided [13.35 to 26.77]
Statistical Analysis 2: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — The effect of TAK-925 was evaluated with a linear mixed effects model appropriate for a 4-period crossover study. The LSM sleep latency for each treatment and the associated standard error and 95% CI was estimated from the model at each time, along with differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p < 0.001, Linear mixed effect model; LSM difference = 24.35, 95% CI 2-sided [17.64 to 31.06]
Statistical Analysis 3: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Linear mixed effects model; LSM Difference = 19.89, 95% CI 2-sided [13.30 to 26.49]

2. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-925 and Its Metabolites M-I and M-II
Time Frame: Day 1 pre-dose and at multiple time points (up to 9 hours) post-dose
Population: The pharmacokinetic (PK) analysis set consisted of all participants who received at least 1 dose of study drug and have at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | TAK-925 44 mg | TAK-925 112 mg
Number analyzed (Participants) | 18 | 18
hour*nanogram per milliliter (h*ng/mL)
  TAK-925 | 940.4 (127.26) | 2303.7 (174.23)
  M-I | 572.0 (196.75) | 1368.3 (489.96)
  M-II | 12.3 (7.91) | 30.7 (19.39)

3. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-925 and Its Metabolites M-I and M-II
Time Frame: Day 1 pre-dose and at multiple time points (up to 9 hours) post-dose
Population: The PK analysis set consisted of all participants who received at least 1 dose of study drug and have at least 1 measurable plasma concentration. The PK analysis set where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TAK-925 44 mg | TAK-925 112 mg
Number analyzed (Participants) | 18 | 18
h*ng/mL
  TAK-925 | 963.7 (134.70) | 2368.7 (185.04)
  M-I | 586.8 (204.08) | 1405.6 (510.25)
  M-II: number analyzed (Participants) | 15 | 18
  M-II | 15.2 (7.38) | 32.0 (20.26)

4. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-925 and Its Metabolites M-I and M-II
Time Frame: Day 1 pre-dose and at multiple time points (up to 9 hours) post-dose
Population: The PK analysis set consisted of all participants who received at least 1 dose of study drug and have at least 1 measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TAK-925 44 mg | TAK-925 112 mg
Number analyzed (Participants) | 18 | 18
nanogram per milliliter (ng/mL)
  TAK-925 | 105.8 (11.74) | 266.0 (40.10)
  M-I | 61.9 (21.41) | 144.7 (55.64)
  M-II | 1.3 (0.88) | 3.2 (2.32)

5. Secondary Outcome: Ceoi: Plasma Concentration Observed at the End of Infusion for TAK-925 and Its Metabolites M-I and M-II
Time Frame: Day 1 pre-dose and at multiple time points (up to 9 hours) post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-925 44 mg | TAK-925 112 mg
Number analyzed (Participants) | 18 | 18
ng/mL
  TAK-925 | 103.4 (14.21) | 253.4 (34.35)
  M-I | 64.0 (21.25) | 151.1 (55.94)
  M-II | 1.5 (0.88) | 3.7 (2.34)

6. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-925 and Its Metabolites M-I and M-II
Time Frame: Day 1 pre-dose and at multiple time points (up to 9 hours) post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | TAK-925 44 mg | TAK-925 112 mg
Number analyzed (Participants) | 18 | 18
hour
  TAK-925 | 9.000 [5.92 to 9.03] | 9.000 [1.07 to 9.02]
  M-I | 9.030 [9 to 9.5] | 9.000 [5.92 to 9.17]
  M-II | 9.170 [9 to 9.5] | 9.000 [5.92 to 9.17]

7. Secondary Outcome: T1/2z: Terminal Disposition Phase Half-life for TAK-925 and Its Metabolites M-I and M-II
Time Frame: Day 1 pre-dose and at multiple time points (up to 9 hours) post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | TAK-925 44 mg | TAK-925 112 mg
Number analyzed (Participants) | 18 | 18
hour
  TAK-925 | 3.134 (0.7064) | 3.252 (0.8597)
  M-I | 2.424 (0.2989) | 2.490 (0.3638)
  M-II: number analyzed (Participants) | 15 | 18
  M-II | 2.235 (0.6945) | 2.516 (0.9660)

8. Secondary Outcome: CL: Total Clearance After Intravenous Administration for TAK-925
Time Frame: Day 1 pre-dose and at multiple time points (up to 9 hours) post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | TAK-925 44 mg | TAK-925 112 mg
Number analyzed (Participants) | 18 | 18
liter per hour (L/h) | 46.4 (5.98) | 47.6 (3.56)

9. Secondary Outcome: Vz: Volume of Distribution During the Terminal Disposition Phase After Intravenous Administration for TAK-925
Time Frame: Day 1 pre-dose and at multiple time points (up to 9 hours) post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | TAK-925 44 mg | TAK-925 112 mg
Number analyzed (Participants) | 18 | 18
liter | 207.4 (41.51) | 223.1 (61.20)

10. Secondary Outcome: Vss: Volume of Distribution at Steady State After Intravenous Administration for TAK-925
Time Frame: Day 1 pre-dose and at multiple time points (up to 9 hours) post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | TAK-925 44 mg | TAK-925 112 mg
Number analyzed (Participants) | 18 | 18
liter | 106.7 (18.90) | 112.5 (25.33)

11. Secondary Outcome: Sleepiness on KSS
Description: The KSS scale measures the subjective level of sleepiness at a particular time during the day. On this scale participants indicate which level best reflects the psycho-physical state experienced in the last 10 minutes. The KSS is a 9-item Likert-type rating scale for assessing subjective sleepiness, where 1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep). Lower score indicates more alertness.
Time Frame: Day 1: 14, 10, 6, 2 hours pre-infusion; 2.75, 4.75, 6.75. 8.75 hours post-infusion start; 1.75 hours post-infusion end
Population: The PD analysis set consisted of all participants who received at least 1 dose of study drug and have at least 1 evaluable postdose PD endpoint derived from the MWT, PSG, KSS, or CCBT. The PD analysis set where data at specified time points was available.
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Groups:
- Placebo: Placebo, once on Day 1 of Intervention Periods 1 to 4.
- Modafinil 300 mg: Modafinil 300 mg, tablet, orally, once on Day 1 of Intervention Periods 1 to 4.
Arm/Group | Placebo | TAK-925 44 mg | TAK-925 112 mg | Modafinil 300 mg
Number analyzed (Participants) | 20 | 18 | 18 | 19
unit on a scale
  14 hours pre-infusion | 3.05 (0.320) | 2.85 (0.339) | 3.29 (0.339) | 2.79 (0.328)
  10 hours pre-infusion | 2.50 (0.283) | 2.79 (0.300) | 2.51 (0.300) | 2.32 (0.291)
  6 hours pre-infusion | 2.80 (0.294) | 2.79 (0.312) | 2.51 (0.312) | 2.58 (0.302)
  2 hours pre-infusion | 3.90 (0.403) | 4.01 (0.426) | 3.46 (0.426) | 3.32 (0.414)
  2.75 hours post -infusion start | 6.85 (0.405) | 4.85 (0.429) | 3.24 (0.429) | 3.69 (0.416)
  4.75 hours post-infusion start | 8.15 (0.376) | 6.46 (0.397) | 3.85 (0.397) | 4.32 (0.386)
  6.75 hours post-infusion start | 8.50 (0.317) | 7.79 (0.336) | 5.18 (0.336) | 5.79 (0.326)
  8.75 hours post-infusion start: number analyzed (Participants) | 19 | 18 | 18 | 19
  8.75 hours post-infusion start | 8.33 (0.325) | 8.07 (0.340) | 6.07 (0.340) | 6.69 (0.330)
  1.75 hours post-infusion end | 8.15 (0.294) | 8.46 (0.312) | 8.01 (0.312) | 7.16 (0.302)
Statistical Analysis 1: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — 14 hours pre-infusion: A linear mixed effect models was performed for all observed KSS parameters at scheduled time points. The LSM sleepless scale for each treatment and the associated standard error and 95% CI was estimated from the model at each time point, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.664, Linear mixed effect model; LSM difference = -0.20, 95% CI 2-sided [-1.13 to 0.73]
Statistical Analysis 2: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.605, Linear mixed effect model; LSM difference = 0.24, 95% CI 2-sided [-0.69 to 1.17]
Statistical Analysis 3: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.574, Linear mixed effect model; LSM difference = -0.26, 95% CI 2-sided [-1.17 to 0.66]
Statistical Analysis 4: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — 10 hours pre-infusion: A linear mixed effect models was performed for all observed KSS parameters at scheduled time points. The LSM sleepless scale for each treatment and the associated standard error and 95% CI was estimated from the model at each time point, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.483, Linear mixed effect model; LSM difference = 0.29, 95% CI 2-sided [-0.53 to 1.11]
Statistical Analysis 5: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 11, analysis 4]; p = 0.972, Linear mixed effect model; LSM difference = 0.01, 95% CI 2-sided [-0.81 to 0.84]
Statistical Analysis 6: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 11, analysis 4]; p = 0.654, Linear mixed effect model; LSM difference = -0.18, 95% CI 2-sided [-0.99 to 0.63]
Statistical Analysis 7: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — 6 hours pre-infusion: A linear mixed effect models was performed for all observed KSS parameters at scheduled time points. The LSM sleepless scale for each treatment and the associated standard error and 95% CI was estimated from the model at each time point, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.984, Linear mixed effect model; LSM difference = -0.01, 95% CI 2-sided [-0.86 to 0.85]
Statistical Analysis 8: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 11, analysis 7]; p = 0.508, Linear mixed effect model; LSM difference = -0.29, 95% CI 2-sided [-1.14 to 0.57]
Statistical Analysis 9: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 11, analysis 7]; p = 0.605, Linear mixed effect model; LSM difference = -0.22, 95% CI 2-sided [-1.06 to 0.62]
Statistical Analysis 10: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — 2 hours pre-infusion: A linear mixed effect models was performed for all observed KSS parameters at scheduled time points. The LSM sleepless scale for each treatment and the associated standard error and 95% CI was estimated from the model at each time point, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.847, Linear mixed effect model; LSM difference = 0.11, 95% CI 2-sided [-1.06 to 1.29]
Statistical Analysis 11: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 11, analysis 10]; p = 0.455, Linear mixed effect model; LSM difference = -0.44, 95% CI 2-sided [-1.61 to 0.73]
Statistical Analysis 12: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 11, analysis 10]; p = 0.317, Linear mixed effect model; LSM difference = -0.58, 95% CI 2-sided [-1.74 to 0.57]
Statistical Analysis 13: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — 2.75 hours post-infusion start: A linear mixed effect models was performed for all observed KSS parameters at scheduled time points. The LSM sleepless scale for each treatment and the associated standard error and 95% CI was estimated from the model at each time point, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.001, Linear mixed effect model; LSM difference = -2.00, 95% CI 2-sided [-3.18 to -0.83]
Statistical Analysis 14: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 11, analysis 13]; p < 0.001, Linear mixed effect model; LSM difference = -3.61, 95% CI 2-sided [-4.79 to -2.44]
Statistical Analysis 15: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 11, analysis 13]; p < 0.001, Linear mixed effect model; LSM difference = -3.16, 95% CI 2-sided [-4.32 to -2.01]
Statistical Analysis 16: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — 4.75 hours post-infusion start: A linear mixed effect models was performed for all observed KSS parameters at scheduled time points. The LSM sleepless scale for each treatment and the associated standard error and 95% CI was estimated from the model at each time point, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.003, Linear mixed effect model; LSM difference = -1.69, 95% CI 2-sided [-2.78 to -0.60]
Statistical Analysis 17: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 11, analysis 16]; p < 0.001, Linear mixed effect model; LSM difference = -4.30, 95% CI 2-sided [-5.39 to -3.21]
Statistical Analysis 18: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 11, analysis 16]; p < 0.001, Linear mixed effect model; LSM difference = -3.83, 95% CI 2-sided [-4.91 to -2.76]
Statistical Analysis 19: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — 6.75 hours post-infusion start: A linear mixed effect models was performed for all observed KSS parameters at scheduled time points. The LSM sleepless scale for each treatment and the associated standard error and 95% CI was estimated from the model at each time point, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.130, Linear mixed effect model; LSM difference = -0.71, 95% CI 2-sided [-1.63 to 0.21]
Statistical Analysis 20: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 11, analysis 19]; p < 0.001, Linear mixed effect model; LSM difference = -3.32, 95% CI 2-sided [-4.24 to -2.40]
Statistical Analysis 21: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 11, analysis 19]; p < 0.001, Linear mixed effect model; LSM difference = -2.71, 95% CI 2-sided [-3.62 to -1.80]
Statistical Analysis 22: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — 8.75 hours post-infusion start: A linear mixed effect models was performed for all observed KSS parameters at scheduled time points. The LSM sleepless scale for each treatment and the associated standard error and 95% CI was estimated from the model at each time point, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.577, Linear mixed effect model; LSM difference = -0.26, 95% CI 2-sided [-1.20 to 0.68]
Statistical Analysis 23: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 11, analysis 22]; p < 0.001, Linear mixed effect model; LSM difference = -2.26, 95% CI 2-sided [-3.20 to -1.32]
Statistical Analysis 24: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 11, analysis 22]; p < 0.001, Linear mixed effect model; LSM difference = -1.65, 95% CI 2-sided [-2.57 to -0.72]
Statistical Analysis 25: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — 1.75 hours post-infusion end: A linear mixed effect models was performed for all observed KSS parameters at scheduled time points. The LSM sleepless scale for each treatment and the associated standard error and 95% CI was estimated from the model at each time point, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.475, Linear mixed effect model; LSM difference = 0.31, 95% CI 2-sided [-0.55 to 1.16]
Statistical Analysis 26: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 11, analysis 25]; p = 0.753, Linear mixed effect model; LSM difference = -0.14, 95% CI 2-sided [-0.99 to 0.72]
Statistical Analysis 27: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 11, analysis 25]; p = 0.022, Linear mixed effect model; LSM difference = -0.99, 95% CI 2-sided [-1.83 to -0.15]

12. Primary Outcome: Latency to Sleep Onset on MWT at 4 Hours Post-infusion Start
Description: as for outcome 1
Time Frame: Day 1: 4 hours post-infusion start
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: minute
Arm/Group | Placebo | TAK-925 44 mg | TAK-925 112 mg | Modafinil 300 mg
Number analyzed (Participants) | 20 | 18 | 18 | 19
minute | 9.10 (2.186) | 32.04 (2.320) | 40.05 (2.320) | 35.60 (2.246)
Statistical Analysis 1: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Linear mixed effect model; LSM difference = 22.94, 95% CI 2-sided [16.58 to 29.30]
Statistical Analysis 2: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Linear mixed effects model; LSM difference = 30.95, 95% CI 2-sided [24.59 to 37.31]
Statistical Analysis 3: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Linear mixed effect model; LSM difference = 26.50, 95% CI 2-sided [20.24 to 32.75]

13. Primary Outcome: Latency to Sleep Onset on MWT at 6 Hours Post-infusion Start
Description: as for outcome 1
Time Frame: Day 1: 6 hours post-infusion start
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: minute
Arm/Group | Placebo | TAK-925 44 mg | TAK-925 112 mg | Modafinil 300 mg
Number analyzed (Participants) | 20 | 18 | 18 | 19
minute | 6.15 (2.589) | 20.71 (2.742) | 38.36 (2.742) | 31.89 (2.659)
Statistical Analysis 1: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Linear mixed effect model; LSM difference = 14.56, 95% CI 2-sided [7.04 to 22.08]
Statistical Analysis 2: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Linear mixed effect model; LSM difference = 32.21, 95% CI 2-sided [24.68 to 39.73]
Statistical Analysis 3: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Linear mixed effect model; LSM difference = 25.74, 95% CI 2-sided [18.33 to 33.14]

14. Primary Outcome: Latency to Sleep Onset on MWT at 8 Hours Post-infusion Start
Description: as for outcome 1
Time Frame: Day 1: 8 hours post-infusion start
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: minute
Arm/Group | Placebo | TAK-925 44 mg | TAK-925 112 mg | Modafinil 300 mg
Number analyzed (Participants) | 20 | 18 | 18 | 19
minute | 3.53 (2.146) | 13.13 (2.279) | 36.86 (2.279) | 20.44 (2.206)
Statistical Analysis 1: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.003, Linear mixed effect model; LSM difference = 9.60, 95% CI 2-sided [3.35 to 15.85]
Statistical Analysis 2: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Linear mixed effect model; LSM difference = 33.33, 95% CI 2-sided [27.08 to 39.58]
Statistical Analysis 3: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Linear mixed effect model; LSM difference = 16.91, 95% CI 2-sided [10.77 to 23.06]

15. Primary Outcome: Latency to Sleep Onset on MWT at 1 Hour Post-end of Infusion
Description: as for outcome 1
Time Frame: Day 1: 1 hour post-end of infusion
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: minute
Arm/Group | Placebo | TAK-925 44 mg | TAK-925 112 mg | Modafinil 300 mg
Number analyzed (Participants) | 20 | 18 | 18 | 19
minute | 4.65 (2.109) | 2.49 (2.241) | 2.36 (2.241) | 21.42 (2.168)
Statistical Analysis 1: Comparison: Placebo vs TAK-925 44 mg; Test type: Superiority — An analysis of variance (ANOVA) model was used to evaluate the 1 hour post the end of infusion MWT. The LSM sleep latency for each treatment and the associated standard error and 95% CI were estimated from the model, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.436, ANOVA; LSM difference = -2.16, 95% CI 2-sided [-7.68 to 3.36]
Statistical Analysis 2: Comparison: Placebo vs TAK-925 112 mg; Test type: Superiority — ANOVA model was used to evaluate the 1 hour post the end of infusion MWT. The LSM sleep latency for each treatment and the associated standard error and 95% CI were estimated from the model, along with the differences between active treatments and placebo, and associated standard errors, 95% CIs, and p-values; p = 0.409, ANOVA; LSM difference = -2.29, 95% CI 2-sided [-7.81 to 3.23]
Statistical Analysis 3: Comparison: Placebo vs Modafinil 300 mg; Test type: Superiority — [test comment as in outcome 15, analysis 2]; p < 0.001, ANOVA; LSM difference = 16.77, 95% CI 2-sided [11.37 to 22.18]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events (AE) that started after the first dose of study drug and no more than 7 days after the last dose of study drug in Treatment Period 4 (Day 1 up to Day 36)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-925 44 mg | TAK-925 112 mg | Modafinil 300 mg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 4/20 | 5/18 | 11/18 | 11/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | TAK-925 44 mg (N=18) | TAK-925 112 mg (N=18) | Modafinil 300 mg (N=19)
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Discomfort (General disorders) | 0 | 0 | 1 | 0
Feeling jittery (General disorders) | 0 | 0 | 1 | 0
Feeling of relaxation (General disorders) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Hypervigilance (Psychiatric disorders) | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 3 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 1
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT03522506/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT03522506/SAP_001.pdf